CLINICAL TRIAL: NCT04653064
Title: Placebo Effects on Anxiety and Pain
Brief Title: The Warmth, Anticipation, Sensation, Aversion, and Body-part Imaging Study
Acronym: WASABI
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Trustees of Dartmouth College (Other)
Responsible Party: Principal Investigator, Tor Wager, Diana L. Taylor Distinguished Professor, Trustees of Dartmouth College
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: 230135
Record Dates: First submitted 2020-11-16; First posted 2020-12-04 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo Cream first (Experimental): Each participant will undergo thermal pain tasks after being administered a "treatment" cream to one of eight body sites.
  Interventions: Behavioral: Placebo Cream; Behavioral: Control Cream
- Control Cream first (Experimental): Each participant will undergo thermal pain tasks after being administered a "control" cream to one of eight body sites.
  Interventions: Behavioral: Placebo Cream; Behavioral: Control Cream

INTERVENTIONS:
Behavioral: Placebo Cream — Approximately 1 teaspoon of exfoliating skin scrub delivered approximately 5 minutes prior to pain tasks will coincide with verbal descriptors of the cream as being analgesic.
Behavioral: Control Cream — Approximately 1 teaspoon of exfoliating skin scrub delivered approximately 5 minutes prior to pain tasks will coincide with verbal descriptors of the cream as one of no effect.

SUMMARY:
This functional magnetic-resonance imaging study of the brain will feature a within-subject crossover design to investigate the effects of a placebo cream on painful thermal stimulation rendered upon eight body sites. The investigators aim to 1.) improve the understanding of how the brain represents thermal pain responses somatotopically (i.e., across different body-sites) 2.) to test these brain representations with and without the presence of a pain-targeted placebo intervention, and 3.) to examine how these brain representations change prior to vs. during the delivery of thermal pain. They predict that placebo cream will downregulate the intensity of aversive brain activity representations, and to a lesser degree, sensation and somatotopic representations, both prior to and during painful thermal stimulation.

DETAILED DESCRIPTION:
Background:

Pain is a significant problem within and outside of clinical contexts, and understanding the phenomenon is imperative for optimizing patient care and understanding the efficacy of pain treatment. At the same time, pain anxiety handicaps behavior and productivity, impedes the adoption of healthy behaviors and proper healthcare delivery, and is implicated in the development and maintenance of chronic pain disorders.

Pain is commonly perceived as a simplistic attention-capturing stimulus response homeostatic monitoring system that serves a tissue-protective function. Contemporary research, however, promotes a process model of pain that goes beyond simple transmission of a nociceptive signal from a transduced stimulus to include aspects of physiological modulation (e.g., regulatory brain activity from midbrain and brainstem, endogenous and exogenous opioids, and experiential perception (e.g., perceptual brain activity from S1, PFC, thalamus, S2, insula, and thalamus, perceptual exercises such as body vision. Clearly, accurate understanding of pain requires require combining signals across brain regions and networks Our lab, using machine-learning based multivoxel pattern analysis (MVPA) have trained several now widely-used whole-brain neural signatures for pain experience using thermal pain delivery devices (e.g., Neural Pain Signature [NPS]), as well as pain-related processes such as viewing pictures of others in pain (Vicarious Pain Signature [VPS]), and imagining being romantically rejected. Pursuit of this line of work has revealed these signatures are sensitive and specific to the type of pain it was developed for, yet generalizable enough to work in samples and pain modalities it was not developed in. For example, NPS is specific to somatic pain, and rises and falls with levels of somatic pain of many types, including thermal pain, mechanical pain, and electric shock, but does not track vicarious pain.

Our existing signatures do not respond to psychological changes in pain, which is believed to be necessary components for understanding pain hyper- and hypo-algesia as well as the placebo effect. The placebo effect is a powerful demonstration of the effects of the psychological pain context on pain experience. The effect may be directly attributable to emotional and attentional processing. Pain processing shifts from nociceptive somatosensory to emotional during chronification of pain and there is ample evidence that anxiety and stress modulate the amounts of pain reported, the degree of treatment and attention requested, and the degree of pain analgesia experienced upon application of placebo. This evidence suggests that aversive processing of incoming stimuli may play a role in the pain experience. Placebo effects may also simply be somatotopically attention driven, as one previous non fMRI study has suggested.

The basic mechanisms of placebo effects on pain anticipation and pain anxiety, and how they relate to placebo effects on pain, are still unknown. Understanding how each of subcomponents of pain -- theoretically separable as the detection of incoming sensation, aversive experiencing, and somatotopic location -- is affected by a placebo treatment may elucidate important facts about pain. This includes how pain is anticipated, processed, and subsequently regulated, providing insight into the nature of pain anxiety and how information should be delivered to mitigate pain. Such knowledge is essential for enhancing existing therapies and creating more nuanced and targeted ones for debilitating pain-related maladies such as chronic pain disorders, and important therapeutic procedures that may cause pain (e.g., surgical or dental).

Experimental Design:

The first hour of fMRI scanning aims to isolate sensation, aversiveness, and somatotopic subcomponents of pain into individual neural signatures. We will do so by subjecting participants at random to stimulations of painful heat and non-painful warmth on various body sites -- left and right masseter, midline chest, midline trunk, left and right forearm, and left and right upper-calf -- as well as listen to an aversive sound (e.g., scratching chalkboard). Participants will also be asked at various times to follow instructions to imagine themselves feeling intense heat pain at a randomly designated body site.

In the second hour of fMRI scanning, we will examine to what degree the identified isolated subcomponents of sensation, aversiveness, and somatotopy respond to placebo treatment for heat pain (i.e., the application of an inert cream coinciding with either an instruction that the participant will be given "an analgesic cream" relative to "a control cream with no effect").

ELIGIBILITY:
Inclusion Criteria:

* Subject must be a volunteer with a minimum age of 18 years and must be able and willing to provide written informed consent.
* If female, the subject must be non-lactating, not pregnant, and using a reliable contraception method.
* Subject must be able to read and speak English.
* Subject must be able to understand and follow the instructions of the investigator and understand all screening questionnaires.
* Subject must have no current or recent history of pathological pain.
* Subject must have abstained from alcohol and substance use for 48 hours.
* Subject must pass all fMRI screening tests.

Exclusion Criteria:

* If female, pregnancy.
* Inability to tolerate the scanning procedures (e.g., claustrophobia).
* Metal in body or prior history working with metal fragments (e.g., as a machinist).
* Inability to tolerate heat pain applied to the forearm.
* Reporting temporary abnormal levels of pain.
* Allergic response to the exfoliating cream.
* Current presence of pain.
* Current or past history of psychoactive substance abuse or dependence.
* Dementias.
* Movement disorders except familial tremor.
* CNS infection.
* CNS vasculitis.
* Inflammatory disease or autoimmune disease.
* CNS demyelinating disease (e.g. multiple sclerosis).
* Space occupying lesions (mass lesions, tumors).
* Congenital CNS abnormality (e.g. cerebral palsy).
* Seizure disorder.
* History of closed head trauma with loss of consciousness.
* History of cerebrovascular disease (stroke, TIAs).
* Abnormal MRI (except changes accounted for by technical factors or UBOs.
* Neuroendocrine disorders (e.g., Cushings disease).
* Uncorrected hypothyroidism or hyperthyroidism.
* Current or past history of cancer.
* Recent history (within two years) of myocardial infarction, severe cardiovascular disease, or currently active cardiovascular disease (e.g. angina, cardiomyopathy).
* Uncontrolled hypertension or hypotension.
* Chronic pain syndromes.
* Chronic fatigue syndromes.
* A history of neurologic disease or neuropathic pain.
* Prior treatment within the last month with any of the following: antidepressants, mood stabilizers, glucocorticoids, opiates.
* Prior treatment with any of the following: antipsychotics, isoniazid, centrally active antihypertensive drugs (e.g. clonidine, reserpine).
* Any other contraindications for MRI examination (e.g., metallic implants such as pacemakers, surgical aneurysm clips, or known metal fragments embedded in the body).
* Current treatment for psychiatric disorders including mood, anxiety, substance abuse, attention-deficit/hyperactivity disorder (ADHD), psychosis.
* Neurological disorders (e.g., taking dopamine agonists for Parkinson's) Cardiovascular disease or medication (e.g., taking ACE (angiotensin-converting-enzyme) inhibitors for cardiac remodeling).
* Frequent smoking (> 5 cigarettes / day).
* Frequent alcohol use (> 14 drinks / week).
* Frequent migraines (> 5 / month on average).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2021-03-19 (Actual); Primary Completion 2026-02-26 (Estimated); Study Completion 2026-12-26 (Estimated)

PRIMARY OUTCOMES:
Contrasts of pain valence (i.e., unpleasantness) using the Bartoshuk Labeled Magnitude Scale (LMS) between body sites administered Placebo vs. Control Cream, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  Self-reported pain valence using the LMS ranging from 0-10 (with 0 representing "no pain" and 10 representing "most unlikable pain of any kind experienced".
Contrast of pain intensity using the Bartoshuk Labeled Magnitude Scale (LMS) between body sites administered Placebo vs. Control Cream, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  Self-reported pain intensity using the LMS ranging from 0-10 (with 0 representing "not intense" and 10 representing "most intense pain of any kind experienced".

SECONDARY OUTCOMES:
Contrasts of activation of fMRI aversiveness signatures between trials where Placebo-cream-applied body sites are stimulated vs. trials where Control-cream-applied body sites are stimulated, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  This will be collected with a Siemens 3T PRISMA.
Contrasts of activation of fMRI sensation signatures between trials where Placebo-cream-applied body sites are stimulated vs. trials where Control-cream-applied body sites are stimulated, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  This will be collected with a Siemens 3T PRISMA.
Contrasts of activation of eight fMRI somatotopic signatures between trials where Placebo-cream-applied body sites are stimulated vs. trials where Control-cream-applied body sites are stimulated, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  This will be collected with a Siemens 3T PRISMA. Eight signatures will include left and right masseter, left and right forearm, left and right calf, sternum, and abdomen.

OTHER OUTCOMES:
Contrast of scalar activation of Neurologic Pain Signature between trials where Placebo-cream-applied body sites are stimulated vs. trials where Control-cream-applied body sites are stimulated, both prior to and during pain delivery. | Hour 2 of fMRI scanning, immediately after each pain delivery trial.
  This will be collected with a Siemens 3T PRISMA.

CONTACTS AND LOCATIONS:
Overall Officials: Tor D Wager, PhD, Principal Investigator — Dartmouth College
Locations (1):
- Dartmouth College, Hanover, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
All MRI and behavioral data will be submitted to the NIMH Data Archive (NDA) according to the terms and conditions outlined on their website (https://ndar.nih.gov/contribute_data_sharing_regimen.html ) and with OpenFMRI.
  All training and test data and multivariate models will also be stored in http://neurovault.org/, an open-source neuroimaging data repository that can accommodate single subject images and metadata used for training multivariate models. We have recently built http://neuro-learn.org/, a new open-source platform for training, testing, and comparing brain models using data stored in Neurovault. All of our neural signatures developed in this project will be made freely available to everyone through this platform.
  All scripts developed to analyze data for this project will be made publicly available on Github (https://github.com/canlab/CanlabCore) at the time of publication of primary manuscripts.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: All data will be de-identified prior to sharing. Raw data will be submitted to NDA within one year from the end of data collection or 6 months from the acceptance date of the first primary study manuscript on the full dataset (excluding methods development papers), whichever is later. Analyzed data/maps of statistical results and models accompanying each paper will be submitted to NDA/OpenFMRI when the primary study manuscript is accepted. All data will be shared indefinitely.
Access Criteria: These data would generally be made available to any qualified investigator for neuroimaging studies only including:
  i. Research on any brain phenomenon; ii. Neuroimaging research on non-disease traits (intelligence, behavioral traits); iii. Methods development research.
  The requesting investigator must provide documentation of local IRB approval.
  These data would not be made available to:
  i. Any criminal justice organization, because data may not be used for any criminal justice applications; ii. Any commercial entity, because use of the data is limited to not-for-profit organizations and data may not be used for any commercial purposes.

DOCUMENTS (1):
  • Informed Consent Form (2020-11-25): https://cdn.clinicaltrials.gov/large-docs/64/NCT04653064/ICF_000.pdf